CLINICAL TRIAL: NCT06537739
Title: Influence of Verbal Suggestion on the Therapeutic Effect of the Joint Manipulation of the Lumbar Spine in Patients with Chronic Non-specific Low Back Pain
Brief Title: Influence of Verbal Suggestion on the Therapeutic Effect of the Joint Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Paul II University in Biała Podlaska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JohnPaul2U
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Back Pain
Keywords: Back Pain; Musculoskeletal Manipulations; Nocebo Effect; Placebo Effect
MeSH Terms: conditions — Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: It will be a prospective follow-up study, with a type of message used as a differentiating variable (positive - placebo, negative - nocebo, neutral).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomly assigned to groups. One of the researchers will then give the person a verbal message (dependent on the study group). The physiotherapist performing the joint manipulation will not know which study group a given patient belongs to. The researcher collecting results and performing statistical analysis will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (test intervention + placebo communication) (Experimental): Participants who will undergo the joint manipulation of the lumbar spine region and receive positive communication - placebo.
  Interventions: Other: Lumbar manipulation; Other: Positive communication - placebo
- Group B (test intervention + nocebo communication) (Experimental): Participants who will undergo the joint manipulation of the lumbar spine region and receive negative communication - nocebo.
  Interventions: Other: Lumbar manipulation; Other: Negative communication - nocebo
- Group C (test intervention + neutral communication) (Other): Participants who will undergo the joint manipulation of the lumbar spine region and receive neutral communication.
  Interventions: Other: Lumbar manipulation; Other: Neutral communication

INTERVENTIONS:
Other: Lumbar manipulation — Participant lies in the supine position, a physiotherapist faces the participant's side that will be manipulated. The participant interlocks their fingers behind their neck. Then the physiotherapist turns the participant on their side and performs a short thrust across the participant's pelvis in a posterior and inferior direction. The manipulation will be carried out on the symptomatic side, based on the participant's indication of the painful side. If the participant is unable to indicate the more symptomatic side, the physiotherapist performing the procedure will select the side. If no audible cavitation occurs during the manipulation, the physiotherapist will attempt to manipulate the opposite side. A maximum of 2 attempts per side will be allowed.
Other: Positive communication - placebo — Participants from Group A who will undergo the joint manipulation of the lumbar spine region and receive the following information: "Joint manipulation is a very effective method of treating spinal disorders, which will significantly reduce the low back pain you are experiencing" (positive communication - placebo).
  Arms: Group A (test intervention + placebo communication)
Other: Negative communication - nocebo — Participants form Group B who will undergo the joint manipulation of the lumbar spine region and receive the following information: "Joint manipulation is not an effective method of treating spinal disorders, thus it may temporarily increase the low back pain you are experiencing" (negative communication - nocebo).
  Arms: Group B (test intervention + nocebo communication)
Other: Neutral communication — Participants from Group C who will undergo the joint manipulation of the lumbar spine region and receive the following information: "Joint manipulation has not been verified for its effectiveness in affecting your level of low back pain" (neutral communication).
  Arms: Group C (test intervention + neutral communication)

SUMMARY:
The aim of the study is to evaluate the influence of verbal suggestion on the therapeutic effect of the joint manipulation of the lumbar spine in patients with chronic non-specific low back pain in relation to the pain level, stress, disability, function, sleepiness, tissue temperature and selected blood biochemical markers.

The study participants will be randomly assigned (sealed allocation envelopes) to the following groups:

* Group A (test intervention + placebo communication)
* Group B (test intervention + nocebo communication)
* Group C (test intervention + neutral communication)

The study will mainly consist of the three stages, i.e. before the intervention, immediately after the intervention and 24 hours later.

DETAILED DESCRIPTION:
Pain is complex in nature and is closely related to the secretion of biochemical markers such as cortisol, serotonin and oxytocin. Higher levels of inflammatory markers, cytokines and chemokines have been found in patients with low back pain, which ultimately affect the clinical manifestations observed in the patients.

One of the methods of physiotherapeutic treatment of spinal disorders involving manual diagnostic and therapeutic techniques is manual therapy. In the therapy, among others, joint manipulation techniques are used. However, the mechanisms underlying the effects of the joint manipulation on the body have not been fully explained. Undoubtedly, one of the main mechanisms of action of manual therapy is pain modulation.

In recent years, research has been increasingly focusing on manipulation in a psychological context, including mechanisms of fear-avoidance, pain catastrophizing and kinesiophobia. Furthermore, manipulation can affect immune and endocrine system responses.

One of the significant non-specific effects accompanying any medical procedure is a placebo effect. The way health care professionals discuss, describe and inform patients about characteristic symptoms of a given disease its prevention, diagnosis and treatment, influences the patients' feelings and expectations, which in turn affect their psycho-biological reactions, subjective perception and treatment outcomes.

The appropriate choice of words by clinicians influences patients' responses to medical treatments and procedures, whether active or sham. The way in which information about the outcome of a treatment is communicated to patients can induce the reinforcing effects of a given treatment (placebo) or reverse the clinically proven effects of an active treatment, or even increase its adverse outcomes in the form of a nocebo effect.

The aim of the study is to evaluate the influence of verbal suggestion on the therapeutic effect of the joint manipulation of the lumbar spine in patients with chronic non-specific low back pain in relation to the pain level, stress, disability, function, sleepiness, tissue temperature and selected blood biochemical markers.

Research questions:

1. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to the pain level?
2. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to the stress level?
3. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to the kinesiophobia level?
4. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to the lumbar spine range of motion?
5. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to the disability level?
6. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to sleepiness?
7. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to the tissue temperature of the lumbar spine region?
8. Does the type of verbal suggestion influence the effects of the joint manipulation in relation to the selected blood biochemical markers (cortisol, serotonin and oxytocin)?

The participants will be selected for the study from the group of students from John Paul II University in Biała Podlaska, Poland. The participation in the study will be voluntary.

The study will mainly consist of the three stages, i.e. before the intervention, immediately after the intervention and 24 hours later. Once, before the intervention, a scale will be used for the subjective assessment of the expectations for the treatment outcomes based on the GRoC methodology. The other research tools will be used in two stages: an information questionnaire (before the intervention and 24 hours after the intervention) and a scale for the subjective assessment of the treatment outcomes based on the GRoC methodology (immediately after the intervention and 24 hours later).

ELIGIBILITY:
Inclusion Criteria:

* participants with low back pain lasting more than 3 months,
* participants who have not been taking any non-steroidal anti-inflammatory drugs (NSAIDs) for at least one week prior to the start of the study,
* participants who are not taking any steroid drugs,
* participants who have never had the joint manipulation before,
* participants within the age range of 19-30 years,
* written consent to participate in the study.

Exclusion Criteria:

* participants who are students of physiotherapy,
* participants with a BMI >33,
* participants after a lumbar spine surgery,
* participants who, in the 6 months prior to the start of the study, suffered from a lumbar spine injury,
* participants with diabetes,
* participants with rheumatic diseases,
* participants with endometriosis,
* participants with endocrine diseases,
* participants with acute inflammation in the lumbar spine region and sciatica symptoms.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Before the intervention, immediately after the intervention and 24 hours later
  The participant gives a score expressed in numbers from 0 to 10

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia (TSK) | Before the intervention, immediately after the intervention and 24 hours later
  The 17 item TSK total scores range from 17 to 68, where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
Back Pain Function Scale (BPFS) | Before the intervention, immediately after the intervention and 24 hours later
  In the Back Pain Function Scale (BFPS), the participant assesses twelve actions related to everyday life activity in a scale of 0 to 5. The results fall within a range of 0 to 60 points, whereby the higher the final result, the lower the level of pain.
Perceived Stress Scale (PSS-10) | Before the intervention, immediately after the intervention and 24 hours later
  The scale consists of 10 questions, with answers scored from 0 to 4.
Stress Numerical Rating Scale-11 | Before the intervention, immediately after the intervention and 24 hours later
  The participant gives a score expressed in numbers from 0 to 10.
Roland-Morris Disability Questionnaire (RMDQ) | Before the intervention, immediately after the intervention and 24 hours later
  The participant is asked to tick a statement when it applies to him/her that specific day; this makes it possible to follow changes in time. The end score is the sum of the ticked boxes. The score ranges from 0 (no disability) to 24 (max. disability) depending on the questionnaire used. Roland and Morris omitted describing the various levels of disability (for example, 40%-60% of disability is severe).
Epworth Sleepiness Scale (ESS) | Before the intervention and 24 hours later
  The ESS is a self-administered questionnaire with 8 questions. The participants are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities.
Serological test - cortisol | Before the intervention, immediately after the intervention and 24 hours later
  During the blood collection, the participants will be placed in a sitting position. Before the blood collection, the following information should be reported: susceptibility to bleeding (bleeding diathesis), susceptibility to fainting during blood collection. In order to determine cortisol levels, the laboratory tests (with the use of immunoenzymatic methods (ELISA tests)) will be performed at the Medical Laboratory of the Innovation Research Center of John Paul II University in Biała Podlaska. The result will be expressed in nmol/L.
Serological test - serotonin | Before the intervention, immediately after the intervention and 24 hours later
  During the blood collection, the participants will be placed in a sitting position. Before the blood collection, the following information should be reported: susceptibility to bleeding (bleeding diathesis), susceptibility to fainting during blood collection. In order to determine serotonin levels, the laboratory tests (with the use of immunoenzymatic methods (ELISA tests)) will be performed at the Medical Laboratory of the Innovation Research Center of John Paul II University in Biała Podlaska. The result will be expressed in ng/ml.
Serological test - oxytocin | Before the intervention, immediately after the intervention and 24 hours later
  During the blood collection, the participants will be placed in a sitting position. Before the blood collection, the following information should be reported: susceptibility to bleeding (bleeding diathesis), susceptibility to fainting during blood collection. In order to determine oxytocin levels, the laboratory tests (with the use of immunoenzymatic methods (ELISA tests)) will be performed at the Medical Laboratory of the Innovation Research Center of John Paul II University in Biała Podlaska. The result will be expressed in mU/l.
Tests with a thermal imaging camera (FLIR E54, USA) | Before the intervention, immediately after the intervention and 24 hours later
  The measurement will be taken in the forward lying position at the level of the three segments: L3, L4 and L5, at three points: the spinous process and on its both sides (2 cm from the spinous process laterally) in the area of the extensor muscles of the lumbar spine.The result will be marked in degrees Celsius.
Tests with the Medi-Mouse (Switzerland) | Before the intervention, immediately after the intervention and 24 hours later
  The assessment of the range of motion of the lumbar spine flexion and extension.The result will be expressed in degrees.
The assessment of the pain levels with the Baseline dolorimeter | Before the intervention, immediately after the intervention and 24 hours later
  The measurement will be taken in the forward lying position at the level of the three segments: L3, L4 and L5, at three points: the spinous process and on its both sides (2 cm from the spinous process laterally) in the area of the extensor muscles of the lumbar spine. A participant will be asked to report when they feel pain at an intensity of 1/10, and a researcher will read the pressure on the dolorimeter.
Scale for the subjective assessment of the expectations for the treatment outcomes based on the GRoC methodology | Before the intervention
  15-point Likert scale - from -7 (lowest expectations) to +7 (highest expectations).
Scale for the subjective assessment of the treatment outcomes based on the GRoC methodology | Immediately after the intervention and 24 hours later
  15-point Likert scale - from -7 (significant worsening of symptoms) to +7 (significant improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Zaworski, Ph.D., Study Chair — John Paul II University in Biała Podlaska
Locations (1):
- John Paul II University in Biała Podlaska, Biała Podlaska, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Analytical data will be available through direct contact with the research team and in the publication process as supplementary materials.
Supporting Information: Study Protocol, Analytic Code
Time Frame: From the completion of the research for the next five years.
Access Criteria: Direct contact with the research team.